CLINICAL TRIAL: NCT02240810
Title: PLATINUM Diversity: Outcomes With the Promus PREMIER™ Stent in Women and Minorities (S2326)
Brief Title: PLATINUM Diversity
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2326
Record Dates: First submitted 2014-09-10; First posted 2014-09-16 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Atherosclerosis; Coronary Artery Disease
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PLATINUM Diversity (Overall): PLATINUM Diversity (Overall) population. Test device is Promus PREMIER Everolimus-Eluting Platinum Chromium Coronary Stent System (CSS)
  Interventions: Device: Percutaneous coronary intervention (Promus PREMIER)

INTERVENTIONS:
Device: Percutaneous coronary intervention (Promus PREMIER) — Interventional coronary artery stenting with Promus PREMIER study stent.

SUMMARY:
To compile acute procedural performance and clinical outcomes data for the Promus PREMIER everolimus-eluting coronary stent system in understudied/underserved patient populations including women and minorities.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age
* Patient must sign informed consent form
* Patient has received at least one Promus PREMIER stent
* Patient self-identifies as one or more of the following:

  * Female
  * Black of African Heritage
  * Hispanic/Latino
  * American Indian or Alaska native

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will be selected from clinical locations where subjects are treated with at least one Promus PREMIER everolimus-eluting coronary stent.
Sampling Method: Non-Probability Sample
Enrollment: 1501 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Mehran, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Wayne Batchelor, MD, Principal Investigator — Tallahassee Memorial Hospital
Locations (52):
- United States (52):
  - St Luke's Medical Center, Phoenix, Arizona
  - St Bernards Heart and Vascular, Jonesboro, Arkansas
  - Arkansas Cardiology/Baptist Health Medical Center, Little Rock, Arkansas
  - Central Cardiology Medical Clinic, Bakersfield, California
  - Sharp Chula Vista Medical Center, Chula Vista, California
  - Cardiovascular Consultants Heart Center, Fresno, California
  - UCLA Medical Center, Los Angeles, California
  - Mercy General Hospital, Sacramento, California
  - Capital Research Institute, Washington D.C., District of Columbia
  - Bay Area Cardiology, Brandon, Florida
  - Research Physicians Network Alliance, Hollywood, Florida
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - Charlotte Heart & Vascular, Port Charlotte, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Pepin Heart Hospital and Dr. Kiran C. Patel Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University Hospital, Augusta, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Presence Saint Joseph Medical Center, Joliet, Illinois
  - The Heart Center of Lake County, Merrillville, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cardiovascular Research, LLC (Willis-Knighton), Shreveport, Louisiana
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Delmarva Heart Research Foundation, Salisbury, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - CCA Research, Gulfport, Mississippi
  - North Kansas City Hospital, North Kansas City, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Mount Sinai Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Presbyterian University Hospital, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Palmetto Health, Columbia, South Carolina
  - St. Francis Physician Services Inc., DBA Upstate Cardiology, Greenville, South Carolina
  - Seton Heart Institute, Austin, Texas
  - Methodist Hospital Dallas, Dallas, Texas
  - VA North Texas Health Care System, Dallas, Texas
  - Plaza Medical Center of Forth Worth, Fort Worth, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Christus Santa Rosa Hospital-City Center, New Braunfels, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - Virginia Mason, Seattle, Washington
  - Cardiac Study Center, Tacoma, Washington
  - CAMC Clinical Trials Center, Charleston, West Virginia

REFERENCES:
- [Background] Batchelor W, Kandzari DE, Davis S, Tami L, Wang JC, Othman I, Gigliotti OS, Haghighat A, Singh S, Lopez M, Giugliano G, Horwitz PA, Chandrasekhar J, Underwood P, Thompson CA, Mehran R. Outcomes in Women and Minorities Compared With White Men 1 Year After Everolimus-Eluting Stent Implantation: Insights and Results From the PLATINUM Diversity and PROMUS Element Plus Post-Approval Study Pooled Analysis. JAMA Cardiol. 2017 Dec 1;2(12):1303-1313. doi: 10.1001/jamacardio.2017.3802. PMID 29049508
- [Derived] Epps K, Goel R, Mehran R, Kandzari D, Damluji A, Tehrani B, Sherwood M, Truesdell A, Davis S, Wang JC, Lopez M, Singh S, Underwood P, Allocco D, Batchelor W. Influence of Race/Ethnicity and Sex on Coronary Stent Outcomes in Diabetic Patients. J Soc Cardiovasc Angiogr Interv. 2023 Sep-Oct;2(5):101053. doi: 10.1016/j.jscai.2023.101053. Epub 2023 Aug 4. PMID 38469035
- [Derived] Beerkens FJ, Cao D, Batchelor W, Sartori S, Kandzari DE, Davis S, Tamis L, Wang JC, Othman I, Vogel B, Spirito A, Subramaniam V, Gigliotti OS, Haghighat A, Feng Y, Singh S, Lopez M, Giugliano G, Horwitz PA, Dangas G, Mehran R. Percutaneous Coronary Intervention in Men, Women, and Minorities With a Previous Coronary Artery Bypass Graft Surgery (from the Pooled PLATINUM Diversity and PROMUS Element Plus Registries). Am J Cardiol. 2023 Aug 1;200:204-211. doi: 10.1016/j.amjcard.2023.05.028. Epub 2023 Jun 22. PMID 37354778
- [Derived] Batchelor WB, Damluji AA, Yong C, Fiuzat M, Barnett SD, Kandzari DE, Sherwood MW, Epps KC, Tehrani BN, Allocco DJ, Meredith IT, Lindenfeld J, O'Connor CM, Mehran R. Does study subject diversity influence cardiology research site performance?: Insights from 2 U.S. National Coronary Stent Registries. Am Heart J. 2021 Jun;236:37-48. doi: 10.1016/j.ahj.2021.02.003. Epub 2021 Feb 24. PMID 33636137
- [Derived] Mehran R, Chandrasekhar J, Davis S, Nathan S, Hill R, Hearne S, Vismara V, Pyo R, Gharib E, Hawa Z, Chrysant G, Kandzari D, Underwood P, Allocco DJ, Batchelor W. Impact of Race and Ethnicity on the Clinical and Angiographic Characteristics, Social Determinants of Health, and 1-Year Outcomes After Everolimus-Eluting Coronary Stent Procedures in Women. Circ Cardiovasc Interv. 2019 Apr;12(4):e006918. doi: 10.1161/CIRCINTERVENTIONS.118.006918. PMID 30998393

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PLATINUM Diversity and PROMUS Element Plus US Post Approval study (PE Plus) are two separate studies that have been pooled.
  Only the PLATINUM Diversity subjects (n=1501) are considered to be enrolled in the study. Results for the PROMUS Element Plus study are reported in record NCT01589978
Groups:
- PLATINUM Diversity (Overall): Percutaneous coronary intervention (Promus PREMIER): Interventional coronary artery stenting with Promus PREMIER study stent.
  Overall population.
- PROMUS Element Plus US Post Approval Study: PROMUS Element Plus US Post Approval Study
Period: Overall Study
Arm/Group | PLATINUM Diversity (Overall) | PROMUS Element Plus US Post Approval Study
Started | 1501 | 2681 (correct typo)
Completed | 1441 | 2621
Not Completed | 60 | 60

BASELINE CHARACTERISTICS:
Groups:
- PROMUS Element Plus US Post Approval Study (Overall): PROMUS Element Plus US Post Approval Study
  NOTE: Results for the PROMUS Element Plus study are reported in record NCT01589978
- Total: Total of all reporting groups
Arm/Group | PLATINUM Diversity (Overall) | PROMUS Element Plus US Post Approval Study (Overall) | Total
Number analyzed (Participants) | 1501 | 2681 | 4182
Age, Customized [Count of Participants; unit: Participants]
  18 Years and Older | 1501 | 2681 | 4182
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1057 | 807 | 1864
  Male | 444 | 1874 | 2318
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — NOTE: Patients were able to self-identify as more than one racial/ethnic category
  Participants
    American Indian or Alaska Native | 28 | 9 | 37
    Asian | 14 | 14 | 28
    Black, of African Heritage | 483 | 189 | 672
    Caucasian | 733 | 2318 | 3051
    Hispanic or Latino | 260 | 95 | 355
    Native Hawaiian or Other Pacific Islander | 2 | 9 | 11
    Other | 13 | 20 | 33
    Not Disclosed | 0 | 37 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1501 | 2681 | 4182
Number of Participants with Current Diabetes Mellitus [Count of Participants; unit: Participants]
  Current Diabetes Mellitus | 676 | 989 | 1665
  Type 1 | 27 | 49 | 76
  Type 2 | 608 | 902 | 1510
  Unknown | 41 | 38 | 79
Number of Participants with History of Hyperlipidemia Requiring Medication [Count of Participants; unit: Participants] | 1107 | 2016 | 3123
Number of Participants with History of Hypertension Requiring Medication [Count of Participants; unit: Participants] | 1275 | 2077 | 3352
Number of Participants with Family History of Coronary Artery Disease (CAD) [Count of Participants; unit: Participants] | 839 | 1625 | 2464
Number of Participants with History of Myocardial Infarction (MI) [Count of Participants; unit: Participants] | 450 | 1409 | 1859
Number of Participants with History of Congestive Heart Failure (CHF) [Count of Participants; unit: Participants] | 215 | 275 | 490
Number of Participants with History of Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants] | 607 | 1159 | 1766
Number of Participants with History of Coronary Artery Bypass Graft (CABG) [Count of Participants; unit: Participants] | 205 | 457 | 662
Number of Participants with History of Renal Disease [Count of Participants; unit: Participants] | 248 | 283 | 531
Number of Participants with History of Peripheral Vascular Disease (PVD) [Count of Participants; unit: Participants] | 175 | 299 | 474
Number of Participants with History of Multivessel Disease [Count of Participants; unit: Participants]
  History of Multivessel Disease | 537 | 1151 | 1688
  2-Vessel | 252 | NA — Not assessed as part of this study | NA — Total not calculated because data are not available (NA) in one or more arms.
  3-Vessel | 285 | NA — Not assessed as part of this study | NA — Total not calculated because data are not available (NA) in one or more arms.
Smoking Status [Count of Participants; unit: Participants]
  Current | 331 | 610 | 941
  Never | 603 | 1021 | 1624
  Previous | 545 | 990 | 1535
  Unknown | 22 | 60 | 82

OUTCOME MEASURES:

1. Primary Outcome: Composite Rate of Death, Myocardial Infarction (MI), and Target Vessel Revascularization (TVR)
Description: A Clinical Events Committee (CEC), independent group of physician experts was used to evaluate all reported cases of death, MI, TVR to determine whether they met the specific protocol definition of the event. It is the CEC adjudicated result that is used in the endpoint analysis. Results for the PROMUS Element Plus study are reported in record NCT01589978
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: the outcome measure is the count of individuals that had a CEC event within 365 days post-procedure. The percentage is calculated based on the count over the denominator (patients who have had any CEC events within 365 days post-procedure or who were event-free with the last follow-up at least 335 days post-procedure).
Measure: Count of Participants; unit: Participants
Groups:
- Caucasian Males - PROMUS Element Plus US Post Approval Study: Caucasian males enrolled in the PROMUS Element Plus US Post Approval Study
- Females - PLATINUM Diversity and PE+: All females enrolled in both the PLATINUM Diversity study and PROMUS Element Plus US Post Approval Study.
- Minorities - PLATINUM Diversity and PE+: All minorities enrolled in both the PLATINUM Diversity study and PROMUS Element Plus US Post Approval Study
Arm/Group | PLATINUM Diversity (Overall) | Caucasian Males - PROMUS Element Plus US Post Approval Study | Females - PLATINUM Diversity and PE+ | Minorities - PLATINUM Diversity and PE+
Number analyzed (Participants) | 1479 | 1569 | 1808 | 1029
Participants | 128 | 120 | 155 | 99

2. Secondary Outcome: Death
Description: A Clinical Events Committee (CEC), independent group of physician experts was used to evaluate all reported cases of death to determine whether they met the specific protocol definition of the event. It is the CEC adjudicated result that is used in the endpoint analysis. Results for the PROMUS Element Plus study are reported in record NCT01589978
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PLATINUM Diversity (Overall) | Caucasian Males - PROMUS Element Plus US Post Approval Study | Females - PLATINUM Diversity and PE+ | Minorities - PLATINUM Diversity and PE+
Number analyzed (Participants) | 1479 | 1569 | 1808 | 1029
Participants | 60 | 35 | 62 | 38

3. Secondary Outcome: Myocardial Infarction (MI)
Description: A Clinical Events Committee (CEC), independent group of physician experts was used to evaluate all reported cases of MI to determine whether they met the specific protocol definition of the event. It is the CEC adjudicated result that is used in the endpoint analysis. Results for the PROMUS Element Plus study are reported in record NCT01589978
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PLATINUM Diversity (Overall) | Caucasian Males - PROMUS Element Plus US Post Approval Study | Females - PLATINUM Diversity and PE+ | Minorities - PLATINUM Diversity and PE+
Number analyzed (Participants) | 1479 | 1569 | 1808 | 1029
Participants | 38 | 17 | 34 | 32

4. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: A Clinical Events Committee (CEC), independent group of physician experts was used to evaluate all reported cases of TVR to determine whether they met the specific protocol definition of the event. It is the CEC adjudicated result that is used in the endpoint analysis. Results for the PROMUS Element Plus study are reported in record NCT01589978
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PLATINUM Diversity (Overall) | Caucasian Males - PROMUS Element Plus US Post Approval Study | Females - PLATINUM Diversity and PE+ | Minorities - PLATINUM Diversity and PE+
Number analyzed (Participants) | 1479 | 1569 | 1808 | 1029
Participants | 58 | 86 | 84 | 56

ADVERSE EVENTS:
Time Frame: 1 year
Description: Overall adverse event data were only analyzed for the PLATINUM Diversity Study. Adverse events for the PROMUS Element Plus study are reported in record NCT01589978.
  Multiple Serious Adverse Events may be experienced by the same study Subjects. The total number of participants affected by all adverse events will not be consistent with Total.
  Adverse Events were assessed at each scheduled study follow-up with participants.
Groups:
- PLATINUM Diversity (Overall): Percutaneous coronary intervention (Promus PREMIER): Interventional coronary artery stenting with Promus PREMIER study stent.
  Overall adverse event data were only analyzed for the PLATINUM Diversity Study. Adverse events for the PROMUS Element Plus study are reported in record NCT01589978.
Arm/Group | PLATINUM Diversity (Overall)
All-Cause Mortality (participants affected / at risk) | 60/1501
Serious Adverse Events (participants affected / at risk) | 154/1501
Other Adverse Events (participants affected / at risk) | 26/1501
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLATINUM Diversity (Overall) (N=1501)
Acute myocardial infarction (Cardiac disorders) | 42 (49) — Multiple Serious Adverse Events may be experienced by the same study Subjects. The total number of participants affected by all adverse events will not be consistent with Total.
Myocardial infarction (Cardiac disorders) | 24 (26)
Coronary artery thrombosis (Cardiac disorders) | 16 (17)
Angina pectoris (Cardiac disorders) | 10 (10)
Coronary artery dissection (Cardiac disorders) | 9 (9)
Cardiac arrest (Cardiac disorders) | 8 (8)
Angina unstable (Cardiac disorders) | 8 (8)
Cardio-respiratory arrest (Cardiac disorders) | 6 (6)
Acute coronary syndrome (Cardiac disorders) | 3 (3)
Cardiac failure (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Electromechanical dissociation (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1)
Postinfarction angina (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 12 (14)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 3 (3)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 2 (2)
Death (General disorders) | 6 (6)
Drowning (General disorders) | 1 (1)
Troponin increased (Investigations) | 3 (3)
Blood creatine phosphokinase MB increased (Investigations) | 2 (2)
Cardiac enzymes increased (Investigations) | 1 (1)
Troponin I increased (Investigations) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Septic shock (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Aortic intramural haematoma (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLATINUM Diversity (Overall) (N=1501)
Myocardial infarction (Cardiac disorders) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less